CLINICAL TRIAL: NCT06771856
Title: Time to Step Up to Stepped Care: A Novel Strategy for Cognitive Behavioral Therapy for Insomnia in Chronic Spinal Pain - a Randomized Controlled Trial
Brief Title: Time to Step Up to Stepped Care: A Novel Strategy for Cognitive Behavioral Therapy for Insomnia in Chronic Spinal Pain
Acronym: StepUp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Malfliet Anneleen, Senior Postdoctoral Researcher, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24408_StepUpStudy; 1251225N (Other Grant/Funding Number: Research Foundation Flanders)
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Chronic Spinal Pain
Keywords: insomnia; stepped care; cognitive behavioral therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: To examine the research aims, a three-arm RCT in people with CSP will be used to compare stepped care CBT-i, standard CBT-i, and a usual group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stepped Care CBTi (Experimental): Stepped Care Cognitive Behavioral Therapy for Insomnia (CBTi). The stepped care approach in CBTi entails a two-step approach. Participants in this group all receive an initial entry level session of 1 hour delivered by a trained physiotherapist. Whether or not they are afterwards referred to the second step (standard care CBTi) depends on their remission status.
  Interventions: Behavioral: Standard Care CBTi; Behavioral: Stepped Care CBTi
- Standard Care CBTi (Active Comparator): Standard Care CBTi will take 10 weeks, during which the participant will have access to an online platform and will have and 2 online face-to-face talks with a certified psychologist. For the online lessons, a validated and effective online intervention will be used. The construction of this online intervention was based on self-help materials, research of the literature, and pa-tient interviews. Standard Care CBTi consists of weekly online webinars and/or exercises and incorporates elements commonly used in face-to-face CBTi. The 10-week program covers the follow-ing topics: the sleep-wake system, how sleep problems arise, bed restriction, reprogram the internal clock, daily habits, stress system, etc. The intervention is supported by online coaching: at two specific time points (around week 3 and week 8) the therapist and participant will have a face-to-face online meeting.
  Interventions: Behavioral: Standard Care CBTi
- Usual Care group (No Intervention): In the usual care group, participants will be asked to continue as usual regarding their sleep behavior and pain-related medical use. They can follow regular care for their pain- and/or sleep problem as recommended by their general practitioner. Their medical use and behavior will be monitored. Once data collection has ended in a usual care participant (i.e., at 12 months follow-up), they are offered a Standard Care CBTi intervention.

INTERVENTIONS:
Behavioral: Standard Care CBTi — Standard Care CBTi will take 10 weeks, during which the participant will receive 5 online les-sons and 3 online face-to-face talks with the therapist. The construction of the online intervention was based on self-help materials, research of the literature, and patient interviews. It consists of 5 online les-sons and incorporates elements commonly used in face-to-face CBTi. The 5 online lessons, one introduced every second week, cover the following topics: Education, stimulus control, sleep restriction, relaxation, cognitions. The intervention is supported by online coaching, with feedback aimed at reviewing exercis-es, clarifying information, and motivating patients to continue the course and make necessary behavioral changes.
  Arms: Standard Care CBTi; Stepped Care CBTi
Behavioral: Stepped Care CBTi — The stepped care approach in CBTi entails a two-step approach. Participants in this group all receive an initial entry level session of 1 hour delivered by a trained physiotherapist. Step 1: The "entry level" in this stepped care approach will imply a single, 1-hour long session, administered by a physiotherapist. This single session will cover: 1) education on sleep, sleep pressure, circadian rhythms; 2) introducing entry-level CBT-i principles (e.g., optimizing sleep environment, pre-bedtime food and beverage consumption) 3) pinpointing 2 to 3 of the most relevant strategies for the participant; and 4) creating an action plan for consistent implementation of these strategies over the next month. One month after 'Step 1' the participants' score on the Insomnia Severity Index (T1) will guide further decision making. Those with ISI scores <12 will enter the follow-up phase immediately. Those with ISI scores ≥12 after step 1 will be referred to standard care CBTi.
  Arms: Stepped Care CBTi

SUMMARY:
Chronic spinal pain (i.e., chronic neck pain and chronic low back pain) are highly prevalent, and are known for their immens personal and socio-economic burden. Chronic spinal pain is impacted by many aspects, and in this story, insomnia plays an important role. Clinical insomnia symptoms are very common in people suffering from chronic spinal pain, and the presence of insomnia is known to aggravate the chronic spinal pain symptoms. While research shows that tackling insomnia in these patients is helpful for these patients, the availability of cognitive behavioral therapy, the golden standard to treat insomnia, is unfortunately extremely limited. Therefore this study aims to investigate whether a stepped care approach to cognitive behavioral therapy is a solution to this problem.

DETAILED DESCRIPTION:
RATIONALE

1. The two-way street of chronic spinal pain (CSP) and insomnia: a bidirectional relationship

   Chronic spinal pain (CSP) is a highly prevalent and pressing health concern, known for its ex-tensive health and socioeconomic burden, incl. prolonged sick-leave, reduced quality of life, and substantial socioeconomic costs. Also, CSP ranks as one of the most prominent causes of years lived with disability worldwide. CSP is a multifaceted problem, and is significantly influ-enced by various factors, among which insomnia plays a pivotal role. Insomnia is, in the absence of other intrinsic sleep disorders and shift work, defined as a sleep dissatisfaction associated with difficulties initiating, maintaining or returning to sleep for >3 days/week for >3 months, with a clear impact on daytime functioning. Clinical insomnia symptoms are very common in peo-ple with CSP, with prevalence rates ranging from 53% up to 90%. Consequently, people with CSP experience detrimental daytime effects, such as memory impairment, work-related issues, and reduced quality of life.

   Insomnia is often considered a result of CSP, yet research findings suggest a bidirectional relation-ship between both. Sleep problems can both trigger and sustain pain, indicating a complex interplay where each can amplify the intensity of the other. Thus, the presence of insomnia can hinder treatment effectiveness in CSP. Moreover, insomnia is also associated with de-creased daily functioning and life satisfaction in this population. Notable, people with chronic pain tend to engage in increased physical activity after one night of better sleep. Hence, target-ing sleep-related issues in people with CSP and comorbid insomnia by offering them an appropri-ate treatment for insomnia (i.e. cognitive behavioral therapy) integrated into pain management is found to enhance treatment effects.
2. Cognitive behavioral therapy for insomnia (CBT-i): Gold Standard Treatment

   Cognitive behavioural therapy for insomnia (CBT-i) is the gold standard treatment for treating insomnia. Over 200 systematic reviews and meta-analyses show evidence for its high long-term, clinically meaningful effectiveness. CBT-i is non-pharmacological and aims to rectify mala-daptive sleep-related beliefs and behaviors, by targeting cognitive and behavioural factors that maintain insomnia with a multicomponent approach, incl. sleep hygiene and restriction, stimulus control, cognitive therapy, and relaxation training. International guidelines recommend CBT-i as first-line treatment for insomnia, and its favorable impact extends to people with chronic pain and comorbid insomnia. Notable, in the context of CSP, an RCT evidences substantial enhancements (moderate to large and clinically meaningful effect sizes) in sleep-related pa-rameters and the impact of pain on daily function.
3. Extremely limited accessibility of CBT-i prevents people from benefiting its efficacy

   The compelling evidence outlined above underscores the importance of integrating CBT-i within pain management. The challenge for CBT-i is no longer to prove its credentials, but to punch its weight, as the extremely limited accessibility of CBT-i hinders patients from both en-gaging in and benefiting from CBT-i. This extremely limited accessibility results from the short-age of licenced CBT-i practitioners, alongside a lack of comprehensive training among primary care providers regarding the identification of sleep-related issues and the appropriate referral for such complaints. Moreover, it is worth noting that the traditional and current usual application of CBT-i necessitates a significant investment of the patient's resources in terms of time, energy, and costs. While the efficacy of CBT-i in people with CSP is undeniably established, it is imperative that future research delves into strategies for mitigating these implementation barriers linked to accessibility. A stepped care model enhances resource efficiency by strategically allo-cating the most expensive human resources to situations where they are most essential, and op-timizes the capacity to effectively treat a larger number of individuals at lower levels of care.
4. Breaking down the barriers: A stepped care CBT-i approach as a promising solution

   To mitigate these challenges of CBT-i access in people with CSP, a stepped care approach offers a solution (fig. 2). This involves providing a step 1 ("entry level") characterized by easy access, minimal therapeutic intensity, least inconvenience for patients, cost-effective, and requir-ing minimal specialist time. An evidence-based approach meeting these criteria, involves replacing sleep-interfering behaviors with sleep-promoting ones through education and behavior change councelling, which can aid sleep initiation and maintenance. Essentially, as step 1 is suitable for dissemination by non-specialists such as nurses, doctors, and physiotherapists, it becomes more accessible for people dealing with insomnia. Moreover, its lower required commit-ment facilitates engagement. The stepped care approach implies that not benefiting sufficiently from the initial "entry level" gives access to step 2: comprehensive, highly effective standard CBT-i.
5. Proof of concept for Stepped Care CBT-i in Chronic Conditions: Transforming Treatment Paradigms

Due to its efficacy, clinical impact, cost-effectiveness and feasibility for many psychological inter-ventions, the stepped care approach is put forward by experts as a promising strategy, which can increase access to high quality interventions. Specifically for insomniacs, uncontrolled studies suggest the effectiveness of stepped care CBT-i with a 69% improvement in sleep efficien-cy. In the context of chronic conditions, an uncontrolled trial (n=51) demonstrated a 45% response (with 41% remitted) to a single session of sleep-related education and behavioral counceling, and subsequent standard CBT-i for the unremitted participants resulted in a 79% response rate and 71% remission. Together with an uncontrolled non-inferiority RCT (n=177) which further corrobo-rated the effectiveness of stepped care CBT-i, this evidence positions stepped care CBT-i as a val-uable and accessible alternative to standard interventions. Looking ahead, the focus of the StepUp project, aligns seamlessly with prevailing expert recommendations. While stepped care CBT-i in CSP awaits empirical validation, a qualitative study in clinicians (n=42) and patients (n=10) supports the feasibility of implementing stepped care in clinical practice. Yet, despite recom-mendations and the prevalence and impact of insomnia in CSP, high-quality controlled trials exploring stepped care CBT-i in this population remain lacking. In summary, these compelling findings not only show the potential benefits of stepped care CBT-i, but also underscore the urgent need to extend this transformative paradigm to the CSP population, as high-quality evidence is lacking.

STUDY OBJECTIVES

In light of the aforementioned considerations, the primary research objective is to examine whether stepped care CBT-i, in comparison to standard CBT-i and a usual care group, leads to a high-er rate of remission from insomnia among people with CSP at 6 months post-treatment (i.e. Pri-mary Endpoint).

Secondary objectives are to assess if stepped care CBT-i, relative to standard CBT-i and a usual care group, yields:

1. Improved cost-effectiveness: Analysing the economic implications and efficiency of stepped-care CBT-i compared to the alternatives.
2. Reduced pain-related and/or sleep-related medication use: Investigating the impact on medica-tion as a key of treatment efficacy.
3. Higher treatment adherence at treatment completion: assessing the levels of patient adher-ence throughout the treatment course

A final secondary aim is to evaluate whether stepped care CBT-i surpasses the usual care group in enhancing sleep quality, pain and physical function among people with CSP.

The overarching hypothesis is that stepped care CBT-i equals or surpasses standard care CBT-i in remission efficacy, with added benefits like reduced medication use, and improved adherence and cost-effectiveness. Additionally, stepped care CBT-i is expected to surpass the usual group in improving sleep quality.

STUDY DESIGN

To examine the research aims, a three-arm RCT in people with CSP will be used to compare stepped care CBT-i, standard CBT-i, and a usual care group. Outcome assessments will take place at baseline, 1 month (T1 = during the intervention period), 3 months (T2 = directly post-treatment), and 9 months (T3 = 6 months follow-up). T1 is the time point where participants in the stepped care group who have not remitted after the entry level (step 1) treatment will continue with receiving comprehensive CBT-I (step 2). T2 is the immediate post-treatment assessments after comprehen-sive CBT-i (both for stepped care CBT-i and the standard CBT-i groups). Participants will be considered treatment responders if their Insomnia Severity Index (ISI) score improves by ≥8 points and will be considered as having remitted if their posttreatment ISI score is <12. Participants ran-domized to the stepped care CBT-i group whose ISI remained ≥12 after step 1 will be referred to step 2.

ELIGIBILITY:
Inclusion Criteria:

Insomniacs (18-65y/o), with an Insomnia Severity Index score ≥15 (i.e., at least moderate insomnia) suffering from CSP, defined as non-specific spinal pain of at least 3 month's duration, currently seeking care for CSP, with a pain severity of ≥3/10 on the Brief Pain Inventory are recruited. In the absence of other intrin-sic sleep disorders and shift work, insomnia is defined as >30 minutes sleep latency and/or minutes awake after sleep onset for >3 days/week for >3 months.

Exclusion Criteria:

Having severe underlying sleep pathology, being pregnant or given birth in the preceding year, suffering from a chronic condition which is currently causing other pain complaints, or suffering from severe psychological or psychiatric dis-eases, dementia or cognitive impairment. Eligible participants are asked not to start new treatments or medication, and continuing the usual non-physical thera-py care (6 weeks prior to and during study participation to obtain a steady state). A sleep-related anamnesis and a polysomnography assessment are performed to determine and exclude severe underlying comorbid sleep disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of remission from insomnia | 6 months post-treatment
  Rate of insomnia remission will be assessed using the Insomnia Severity Index (ISI), a self-report questionnaire assessing the nature, severity, and impact of insomnia. Participants will be considered treatment responders if their Insomnia Severity Index (ISI) score improves by ≥8 points and will be considered as having remitted if their post-treatment ISI score is <12.

SECONDARY OUTCOMES:
Insomnia Severity | Change from baseline to directly post-treatment, 6 months and 12 months follow-up
  Change in insomnia severity will be assessed using the Insomnia Severity Index (ISI), a self-report questionnaire assessing the nature, severity, and impact of insomnia. Each item scored on a Likert scale ranging from 0 (no problem) to 4 (very severe problem) yields a total score, interpreted as: 0-7 = absence of insomnia; 8-14 = sub-threshold insomnia; 15-21 = moderate insomnia; and 22-28 = severe insomnia. The score will be used as a continuous variable in the analysis.
Medical Consumption Questionnaire | At baseline, 6 months follow-up and 12 months follow-up.
  The Medical Consumption Questionnaire (MCQ) is an instrument for measuring medical consumption. The MCQ includes questions related to frequently occurring contacts with health care providers.
Productivity Cost Questionnaire | At baseline, 6 months follow-up and 12 months follow-up.
  The Productivity Cost Questionnaire (PCQ) is a recall questionnaire that collects data related to loss of productivity in paid and unpaid work.
Health-related quality of life | At baseline, 6 months follow-up and 12 months follow-up.
  The EQ-5D is a standardized instrument used to assess five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by assigning a score. From this, a weighted health index can be derived for an individual or a population.
Sleep quality | At baseline, directly post-treatment, at 6 months follow-up and at 12 months follow-up
  The Pittsburg Sleep Quality Index is used to evaluate overall self-reported sleep quality.
Sleepiness | At baseline, directly post-treatment, at 6 months follow-up and at 12 months follow-up
  Self-reported sleepiness is assessed using the Epworth sleepiness scale, which is widely used in the field of sleep medicine as a subjective measure of a patient's sleepiness. The test is a list of eight situations in which the patient rates his/her tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing.
Pain intensity and interference | At baseline, directly post-treatment, at 6 months follow-up and at 12 months follow-up
  The Brief Pain Inventory (BPI) assesses pain severity and pain interference in daily life over the past week.
Quality of Life | At baseline, directly post-treatment, at 6 months follow-up and at 12 months follow-up
  The SF-36 is often used as a measure of a person or population's quality of life. It compris-es 36 questions that cover eight domains of health: 1) Limitations in physical activities be-cause of health problems; 2) Limitations in social activities because of physical or emotion-al problems; 3) Limitations in usual role activities because of physical health problems; 4) Bodily pain; 5) General mental health (psychological distress and well-being); 6) Limitations in usual role activities because of emotional problems; 7) Vitality (energy and fatigue); 8) General health perceptions. The scoring system of the SF36 results into two final scores: one focusing on physical health, and one focusing on mental health.
Symptoms of anxiety and depression | At baseline, directly post-treatment, at 6 months follow-up and at 12 months follow-up
  The Hospital Anxiety and Depression Scale (HADS) is used as an indicative measurement of anxiety and depression.
Fatigue | At baseline, directly post-treatment, at 6 months follow-up and at 12 months follow-up
  The Brugmann Fatigue Scale is used to assess self-reported fatigue severity with a mental fatigue subscale and physical fatigue subscale. The score ranges from 0 to 24 and higher scores indicate a higher subjective level of fatigue.
Treatment adherence | Directly post-treatment
  In the two treatment groups treatment adherence will be questioned using the Treatment Adherence Perception Questionnaire (TAPQ). This is a brief self-report instrument for as-sessing patient perceptions and attitudes regarding their own adherence to medical treat-ment plans. It includes 3 distinct scales: Perceived Behavior, Perceived Benefit, and Per-ceived Burden.
Objective sleep assessment | At baseline, directly post-treatment and at 6 months follow-up
  Participants will undergo a one night polysomnography assessment at home, using the MUSE S headband (InteraXon, Canada - https://choosemuse.com).

OTHER OUTCOMES:
Demographics | Baseline
  Information on age, sex, educational level, employment status, marital status, and ethnici-ty will be collected.
Adverse Events | Directly post-treatment, at 6 months follow-up and at 12 months follow-up
  With each online assessment (except for baseline), adverse events will we questioned in the participants. This will be done using the following question: "What unusual symptoms or medical problems have you experienced since the last round of questionnaires?". Re-ported adverse events will be classified as 'mild' (i.e., mild concentration problems), 'mod-erate' (e.g., fever) or 'serious adverse events' (e.g., death, hospitalization). No moderate or serious adverse events are expected in this trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Given the highly sensitive nature of data, this will not be shared.